CLINICAL TRIAL: NCT00101686
Title: A Randomized, Multi-Center Phase III Trial Of Irinotecan In Combination With Three Different Methods Of Administration Of Fluoropyrimidine: Infusional 5-FU (FOLFIRI), Modified-Bolus 5-FU (Day 1 & 8), And Oral Capecitabine (Day 1-14); With Celecoxib Versus Placebo As First-Line Treatment For Patients With Metastatic Colorectal Cancer Study Amended April 23, 2004 To Include Bevacizumab
Brief Title: Trial Of Irinotecan In Combination With Three Methods Of Administration Of Fluoropyrimidine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPTAIV-0020-411; A5961021
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Modified Bolus 5-FU/LV with Irinotecan (Experimental)
  Interventions: Drug: Modified Bolus 5-FU/LV with Irinotecan
- FOLFIRI + bevacizumab (Experimental)
  Interventions: Drug: FOLFIRI + bevacizumab
- miFL + bevacizumab (Experimental)
  Interventions: Drug: miFL + bevacizumab
- Infusional 5-FU/LV with Irinotecan (Experimental)
  Interventions: Drug: Infusional 5-FU/LV with Irinotecan
- Oral Capecitabine with Irinotecan (Other)
  Interventions: Drug: Oral Capecitabine with Irinotecan

INTERVENTIONS:
Drug: Modified Bolus 5-FU/LV with Irinotecan — Day 1 & 8: Irinotecan (125 mg/m2 IV over 90 minutes), LV (20 mg/m2 IV bolus), 5-FU (500 mg/m2 IV bolus). All chemotherapy cycles repeated every 3 weeks. Celecoxib/placebo treatment will commence on the same day as chemotherapy treatment (i.e. Day 1 of treatment on study). Celecoxib/placebo will be taken at a dose of 400 mg po BID [two times a day] (800 mg/day) and will continue daily without interruption (no rest period for celecoxib/placebo treatment).
  Arms: Modified Bolus 5-FU/LV with Irinotecan
Drug: FOLFIRI + bevacizumab — Day 1 Bevacizumab 5mg/kg IV 90 minutes prior to irinotecan/LV Irinotecan 180 mg/m2 IV 90 minutes Leucovorin 400 mg/m2 IV 2 hours - given with irinotecan without mixing.
  I m m e d i a t e l y f o l l o w e d b y :
  5-FU 400 mg/m2 IV bolus 5-FU 2400 mg/m2 IV Continuous infusion over 46 hours Every 2 weeks
  Amendment 2 Bevacizumab 5mg/kg IV 90 minutes prior to irinotecan/LV Irinotecan 180 mg/m2 IV 90 minutes Leucovorin 400 mg/m2 IV 2 hours - given with irinotecan without mixing.
  I m m e d i a t e l y f o l l o w e d b y :
  5-FU 400 mg/m2 IV bolus 5-FU 2400 mg/m2 IV Continuous infusion over 46 hours Celecoxib/placebo 400 mg BID [two times a day] oral Every 2 weeks
  Arms: FOLFIRI + bevacizumab
Drug: miFL + bevacizumab — Day 1 Bevacizumab 7.5mg/kg IV *over 90 minutes - given prior to irinotecan, 5-FU, and leucovorin Irinotecan 125 mg/m2 IV over 90 minutes Leucovorin 20 mg/m2 IV bolus 5-FU 500 mg/m2 IV bolus Day 8 Irinotecan 125 mg/m2 IV over 90 minutes Leucovorin 20 mg/m2 IV bolus 5-FU 500 mg/m2 IV bolus Every 3 weeks Amendment 2 Day 1 Bevacizumab 7.5mg/kg IV over 90 minutes - given prior to irinotecan, 5-FU, and leucovorin Irinotecan 125 mg/m2 IV over 90 minutes Leucovorin 20 mg/m2 IV bolus 5-FU 500 mg/m2 IV bolus Celecoxib/placebo 400 mg BID [two times a day] oral Day 8 Irinotecan 125 mg/m2 IV over 90 minutes Leucovorin 20 mg/m2 IV bolus 5-FU 500 mg/m2 IV bolus Celecoxib/placebo -- 400 mg po BID [two times a day] continues daily without interruption Every 3 weeks
  Arms: miFL + bevacizumab
Drug: Infusional 5-FU/LV with Irinotecan — Day 1: Irinotecan (180 mg/m2) IV over 90 minutes, LV (racemic mixture 400 mg/m2) over 2 hours during irinotecan infusion but without mixing, immediately followed by 5-FU IV bolus (400 mg/m2) and 5-FU continuous infusion (2400 mg/m2) over 46 hours. FOLFIRI regimen is repeated every 2 weeks. Celecoxib/placebo treatment will commence on the same day at a dose of 400 mg po BID [two times a day](800 mg/day) and will continue daily without interruption (no rest period for celecoxib/placebo treatment).
  Arms: Infusional 5-FU/LV with Irinotecan
Drug: Oral Capecitabine with Irinotecan — Day 1: Irinotecan (250 mg/m2 IV) over 90 minutes; Day 1-14: capecitabine 1000 mg/m2 PO BID [two times a day] (28 single doses). All chemotherapy cycles repeated every 3 weeks. Celecoxib/placebo treatment will commence on the same day as chemotherapy treatment (i.e. Day 1 of treatment on study). Celecoxib/placebo will be taken at a dose of 400 mg po BID (800 mg/day) and will continue daily without interruption (no rest period for celecoxib/placebo treatment).
  Arms: Oral Capecitabine with Irinotecan

SUMMARY:
This study compares in the first study period combination of Irinotecan with three different methods of administration by Fluoropyrimidine. (ie. infusion, bolus and oral). In the second period of study it compares FOLFIRI [a chemotherapy regime that combines bolus irinotecan and leucovorin [LV] with infusional 5-fluorouracil (5-FU)] + bevacizumab and mlFL + bevacizumab. Measures of efficacy and safety will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal cancer (either newly diagnosed or recurrent disease) with evidence of metastatic disease. (Stage IV distant disease)
* Present or past histological documentation of adenocarcinoma of the colon or rectum. The site of the primary lesion must be or have been confirmed endoscopically, radiologically, or surgically to be or have been in the large bowel. Patients with a history of colorectal cancer treated by surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease unless:
* An interval of greater than five years has elapsed between the primary surgery and the development of metastatic disease.
* The primary cancer was a Duke's A or B1.
* Physicians should consider biopsy of lesions to establish the diagnosis of metastatic colorectal cancer in each case if there is substantial clinical ambiguity regarding the nature of source of apparent metastases.

Exclusion Criteria:

* Patients who received any prior systemic anticancer therapy for metastatic colorectal cancer (e.g., chemotherapy, antibody therapy, immunotherapy, gene therapy, vaccine therapy, cytokine therapy, or other experimental agents).
* Patients cannot have concurrent malignancies at study entry.
* Exceptions: Patients with prior non-colorectal malignancies will be eligible if they have been disease-free for ³ 3 years or are deemed at low risk for recurrence by their treating physician (e.g., early stage prostate cancer, melanoma or bladder cancer). Patients with squamous or basal cell carcinoma of the skin or in situ cervical cancer that have been effectively treated are eligible, even if these were diagnosed within 3 years before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2003-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (158):
- United States (126):
  - Pfizer Investigational Site, Birmgingham, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Birmngham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Flagstaff, Arizona
  - Pfizer Investigational Site, Sedona, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Hot Spring, Arkansas
  - Pfizer Investigational Site, Springdale, Arkansas
  - Pfizer Investigational Site, Arroyo Grande, California
  - Pfizer Investigational Site, Fountian Valley, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Los Gatos, California
  - Pfizer Investigational Site, Mission Hills, California
  - Pfizer Investigational Site, Modesto, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Oxnard, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Jose, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Stamford, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Altamonte Springs, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Lauderhill, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Miami Beach, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Tamarac, Florida
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Niles, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Skokie, Illinois
  - Pfizer Investigational Site, Fishers, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Alexandria, Louisiana
  - Pfizer Investigational Site, Shrevport, Louisiana
  - Pfizer Investigational Site, Bangor, Maine
  - Pfizer Investigational Site, Annapolis, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Burlington, Massachusetts
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Burnsville, Minnesota
  - Pfizer Investigational Site, Robbinsdale, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Joplin, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Hooksett, New Hampshire
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Nashua, New Hampshire
  - Pfizer Investigational Site, Summit, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Farmington, New Mexico
  - Pfizer Investigational Site, Santa Fe, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Manhaset, New York
  - Pfizer Investigational Site, Rockville Centre, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Fayetteville, North Carolina
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Hendersonville, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Bartlesville, Oklahoma
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Abington, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Reading, Pennsylvania
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Collierville, Tennessee
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Abilene, Texas
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Bedford, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Denton, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Fredericksburg, Texas
  - Pfizer Investigational Site, Garland, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Lewisville, Texas
  - Pfizer Investigational Site, Longview, Texas
  - Pfizer Investigational Site, McAllen, Texas
  - Pfizer Investigational Site, Mesquite, Texas
  - Pfizer Investigational Site, Midland, Texas
  - Pfizer Investigational Site, New Braunfels, Texas
  - Pfizer Investigational Site, Odessa, Texas
  - Pfizer Investigational Site, Paris, Texas
  - Pfizer Investigational Site, Sherman, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Waco, Texas
  - Pfizer Investigational Site, Webster, Texas
  - Pfizer Investigational Site, Wichita Falls, Texas
  - Pfizer Investigational Site, Colchester, Vermont
  - Pfizer Investigational Site, Fairfax, Virginia
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Roanoke, Virginia
  - Pfizer Investigational Site, Edmonds, Washington
  - Pfizer Investigational Site, Lacy, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Yakima, Washington
  - Pfizer Investigational Site, Glendale, Wisconsin
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Australia (6):
  - Pfizer Investigational Site, Waratah, New South Wales
  - Pfizer Investigational Site, South Brisbane, Queensland
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, Woodville, South Australia
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Frankston, Victoria
- Canada (22):
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Sydney, Nova Scotia
  - Pfizer Investigational Site, Brampton, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Scarborough Village, Ontario
  - Pfizer Investigational Site, Thunder Bay, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Fleurimont, Quebec
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Rimouski, Quebec
  - Pfizer Investigational Site, Regina, Saskatchewan
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- New Zealand (4):
  - Pfizer Investigational Site, Auckland
  - Pfizer Investigational Site, Dunedin
  - Pfizer Investigational Site, Riccarton
  - Pfizer Investigational Site, Wellington

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFIRI + Celecoxib: Irinotecan plus infusional 5-Fluorouracil(5-FU)/Leucovorin(LV) (FOLFIRI) with celecoxib
- FOLFIRI + Placebo: Irinotecan plus infusional 5-FU/LV (FOLFIRI) with placebo
- mIFL + Celecoxib: Modified irinotecan plus bolus 5-FU/LV (mIFL) with celecoxib
- mIFL + Placebo: Modified irinotecan plus bolus 5-FU/LV (mIFL) with placebo
- CapeIRI + Celecoxib: Irinotecan plus capecitabine (CapeIRI) with celecoxib
- CapeIRI + Placebo: Irinotecan plus capecitabine (CapeIRI) with placebo
- Bevacizumab + FOLFIRI + Celecoxib: Bevacizumab + Irinotecan plus infusional 5-FU/LV (FOLFIRI) with celecoxib
- Bevacizumab + FOLFIRI + Placebo: Bevacizumab + Irinotecan plus infusional 5-FU/LV (FOLFIRI) with placebo
- Bevacizumab + mIFL + Celecoxib: Bevacizumab + Modified irinotecan plus bolus 5-FU/LV (mIFL) with celecoxib
- Bevacizumab + mIFL + Placebo: Bevacizumab + Modified irinotecan plus bolus 5-FU/LV (mIFL)with placebo
Period: Overall Study
Arm/Group | FOLFIRI + Celecoxib | FOLFIRI + Placebo | mIFL + Celecoxib | mIFL + Placebo | CapeIRI + Celecoxib | CapeIRI + Placebo | Bevacizumab + FOLFIRI + Celecoxib | Bevacizumab + FOLFIRI + Placebo | Bevacizumab + mIFL + Celecoxib | Bevacizumab + mIFL + Placebo
Started | 71 | 73 | 69 | 72 | 73 | 72 | 27 | 30 | 30 | 30
Received Treatment | 70 | 67 | 67 | 70 | 71 | 70 | 27 | 29 | 30 | 29
Completed | 0 (Patients treated until disease progression.) | 0 (Patients treated until disease progression.) | 0 (Patients treated until disease progression.) | 0 (Patients treated until disease progression.) | 0 (Patients treated until disease progression.) | 0 (Patients treated until disease progression.) | 0 (Patients treated until disease progression.) | 0 (Patients treated until disease progression.) | 0 (Patients treated until disease progression.) | 0 (Patients treated until disease progression.)
Not Completed | 71 | 73 | 69 | 72 | 73 | 72 | 27 | 30 | 30 | 30
Not completed — Progressive Disease | 37 | 28 | 37 | 38 | 28 | 25 | 5 | 7 | 10 | 8
Not completed — initiation other anti-cancer treatment | 4 | 3 | 4 | 3 | 1 | 1 | 2 | 2 | 3 | 3
Not completed — >3 week delay treatment due toxicity | 6 | 2 | 1 | 2 | 7 | 3 | 2 | 1 | 3 | 0
Not completed — unacceptable toxicity | 3 | 9 | 10 | 6 | 16 | 10 | 4 | 2 | 1 | 4
Not completed — Randomized but did not receive treament | 1 | 6 | 2 | 2 | 2 | 2 | 0 | 1 | 0 | 1
Not completed — intercurrent non-cancer related illness | 0 | 0 | 2 | 0 | 1 | 3 | 1 | 0 | 1 | 1
Not completed — Physician Decision | 10 | 13 | 6 | 7 | 8 | 9 | 5 | 5 | 1 | 1
Not completed — Other | 1 | 4 | 1 | 6 | 2 | 12 | 1 | 5 | 3 | 3
Not completed — Withdrawal by Subject | 9 | 8 | 6 | 8 | 8 | 7 | 7 | 7 | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFIRI + Celecoxib | FOLFIRI + Placebo | mIFL + Celecoxib | mIFL + Placebo | CapeIRI + Celecoxib | CapeIRI + Placebo | Bevacizumab + FOLFIRI + Celecoxib | Bevacizumab + FOLFIRI + Placebo | Bevacizumab + mIFL + Celecoxib | Bevacizumab + mIFL + Placebo | Total
Number analyzed (Participants) | 71 | 73 | 69 | 72 | 73 | 72 | 27 | 30 | 30 | 30 | 547
Age Continuous [Median (Full Range); unit: years] | 61.0 [35.0 to 81.0] | 62.0 [31.0 to 87.0] | 61.0 [34.0 to 78.0] | 62.0 [29.0 to 80.0] | 62.0 [20.0 to 78.0] | 62.5 [33.0 to 85.0] | 59.0 [37.0 to 81.0] | 59.5 [32.0 to 80.0] | 61.0 [45.0 to 84.0] | 59.0 [35.0 to 84.0] | 61.0 [20.0 to 87.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 34 | 24 | 29 | 37 | 13 | 14 | 10 | 12 | 225
  Male | 49 | 43 | 35 | 48 | 44 | 35 | 14 | 16 | 20 | 18 | 322

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP) at Primary Completion: FOLFIRI and mIFL
Description: Time to disease progression is defined as the number of months from date of randomization to the date of first documentation of disease progression (PD).
Time Frame: every 6 weeks until disease progression
Population: Intent-to-Treat Population (ITT) - all subjects who were randomized, with study drug assignment designated according to initial randomization, regardless of whether subjects received any study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- FOLFIRI: Irinotecan + infusional 5-FU/LV with celecoxib or placebo
- mIFL: Irinotecan + modified-bolus 5-FU/LV with celecoxib or placebo
Arm/Group | FOLFIRI | mIFL
Number analyzed (Participants) | 144 | 141
months | 8.18 [7.43 to 8.97] | 6.01 [5.52 to 7.03]
Statistical Analysis 1: Comparison: FOLFIRI vs mIFL; Test type: Superiority or Other; p = 0.0152, Log Rank — p-value corresponds to the log-rank test for comparing Kaplan-Meier survival curves; Hazard Ratio (HR) = 1.433, 95% CI [1.09 to 1.89] — Hazard ratio [mIRI:FOLFIRI] is from the Cox Proportional Hazard Model using treatment (FOLFIRI, mIRI, CapeIRI), age (<=70 vs >70), performance status (0 vs 1), aspirin (Yes vs No), celecoxib (Yes or No) as the covariates

2. Secondary Outcome: Time to Progression: FOLFIRI, mIFL and CapeIRI
Description: as for outcome 1
Time Frame: every 6 weeks until disease progression
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CapeIRI: Irinotecan + oral capecitabine with celecoxib or placebo
Arm/Group | FOLFIRI | mIFL | CapeIRI
Number analyzed (Participants) | 144 | 141 | 145
months | 7.62 [7.06 to 8.71] | 5.98 [5.45 to 6.9] | 5.82 [4.60 to 6.9]
Statistical Analysis 1: Comparison: FOLFIRI vs mIFL; Test type: Superiority or Other; p = 0.0042, Log Rank; Hazard Ratio (HR) = 1.512, 95% CI [1.16 to 1.97]
Statistical Analysis 2: Comparison: FOLFIRI vs CapeIRI; Test type: Superiority or Other; p = 0.0156, Log Rank; Hazard Ratio (HR) = 1.368, 95% CI [1.04 to 1.80]
Statistical Analysis 3: Comparison: mIFL vs CapeIRI; Test type: Superiority or Other; p = 0.4659, Log Rank; Hazard Ratio (HR) = 1.057, 95% CI [0.81 to 1.38]

3. Secondary Outcome: Overall Response: FOLFIRI, mIFL and CapeIRI
Description: A subject will be considered achieving an overall response if the subject has a sustained Complete Response (CR) or Partial Response (PR) for at least 4 weeks, confirmed by tumor assessments. (CR: Disappearance of all target lesions. PR: greater than or equal to 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the Pre-treatment sum LD. )
Time Frame: every 6 weeks during chemotherapy until disease progression
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | FOLFIRI | mIFL | CapeIRI
Number analyzed (Participants) | 144 | 141 | 145
participants | 68 | 61 | 56
Statistical Analysis 1: Comparison: FOLFIRI; Test type: Superiority or Other; F-distribution method = 47.2, 95% CI [38.85 to 55.71] — Exact confidence interval for binomial proportion using the F-distribution method (unit: %)
Statistical Analysis 2: Comparison: mIFL; Test type: Superiority or Other; F-distribution method = 43.3, 95% CI [34.95 to 51.86] — Exact confidence interval for binomial proportion using the F-distribution method (unit: %)
Statistical Analysis 3: Comparison: CapeIRI; Test type: Superiority or Other; F-distribution method = 38.6, 95% CI [30.66 to 47.06] — Exact confidence interval for binomial proportion using the F-distribution method (unit: %)
Statistical Analysis 4: Comparison: FOLFIRI vs mIFL; Test type: Superiority or Other; p = 0.4751, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: FOLFIRI vs CapeIRI; Test type: Superiority or Other; p = 0.1591, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: mIFL vs CapeIRI; Test type: Superiority or Other; p = 0.4395, Cochran-Mantel-Haenszel

4. Secondary Outcome: Survival Time: FOLFIRI, mIFL and CapeIRI
Description: Survival time defined as time from date of randomization to date of death. In the absence of confirmation of death, survival time was censored to last date the subject known to be alive.
Time Frame: assessed at least every week during treatment and at least every 3 months during follow-up
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFIRI | mIFL | CapeIRI
Number analyzed (Participants) | 144 | 141 | 145
months | 23.06 [17.87 to 26.55] | 17.64 [14.29 to 23.03] | 18.92 [15.74 to 23.23]
Statistical Analysis 1: Comparison: FOLFIRI vs mIFL; Test type: Superiority or Other; p = 0.0879, Log Rank; Hazard Ratio (HR) = 1.268, 95% CI [0.96 to 1.68]
Statistical Analysis 2: Comparison: FOLFIRI vs CapeIRI; Test type: Superiority or Other; p = 0.2765, Log Rank; Hazard Ratio (HR) = 1.190, 95% CI [0.90 to 1.58]
Statistical Analysis 3: Comparison: mIFL vs CapeIRI; Test type: Superiority or Other; p = 0.9364, Log Rank; Hazard Ratio (HR) = 1.049, 95% CI [0.80 to 1.38]

5. Secondary Outcome: 1 Year Survival: FOLFIRI, mIFL and CapeIRI
Description: Number of patients alive or dead at 1 year. In the absence of confirmation of death, survival time was censored to last date the subject known to be alive.
Time Frame: 1 year from date of randomization
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | FOLFIRI | mIFL | CapeIRI
Number analyzed (Participants) | 144 | 141 | 145
participants
  Alive at 1 year | 101 | 86 | 89
  Dead at 1 year | 34 | 47 | 46
  Censored | 9 | 8 | 10

6. Secondary Outcome: Time to Progression : Celecoxib and Placebo
Description: as for outcome 1
Time Frame: every 6 weeks until disease progression
Population: ITT Population. Celecoxib participants were combined from FOLFIRI, mIRI, and Capecitabine treatments (not bevacizumab); Placebo participants were combined from FOLFIRI, mIRI, and Capecitabine treatments (not bevacizumab).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Celecoxib: All patients treated with celecoxib: combined patients treated with FOLFIRI+ celecoxib, mIRI+ celecoxib, CapeIRI+ celecoxib
- Placebo: All patients treated with placebo: combined patients treated with FOLFIRI+placebo, mIRI+placebo, CapeIRI+placebo
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 213 | 217
months | 6.64 [5.68 to 7.39] | 6.70 [6.01 to 7.26]
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.7163, Log Rank; Hazard Ratio (HR) = 1.068, 95% CI [0.86 to 1.33]

7. Secondary Outcome: Overall Response: Celecoxib and Placebo
Description: A subject will be considered achieving an overall response if the subject has a sustained CR or PR for at least 4 weeks, confirmed by tumor assessments. (Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): ≥ 30% decrease in the sum of the LD of target lesions, taking as reference the Pre-treatment sum LD. )
Time Frame: every 6 weeks during chemotherapy until disease progression
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 213 | 217
participants | 84 | 101
Statistical Analysis 1: Comparison: Celecoxib; Test type: Superiority or Other; F-distribution method = 39.4, 95% CI [32.83 to 46.34] — confidence interval for binomial proportion using the F-distribution method (unit: %)
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; F-distribution method = 46.5, 95% CI [39.76 to 53.42] — confidence interval for binomial proportion using the F-distribution method (unit: %)
Statistical Analysis 3: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.1559, Cochran-Mantel-Haenszel

8. Secondary Outcome: Survival Time: Celecoxib and Placebo
Description: as for outcome 4
Time Frame: assessed at least every week during treatment and at least every 3 months during follow-up
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 213 | 217
months | 21.06 [16.92 to 24.28] | 18.83 [16.26 to 22.93]
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.5316, Log Rank; Hazard Ratio (HR) = 1.080, 95% CI [0.86 to 1.36]

9. Secondary Outcome: Time to Progression: Bevacizumab With FOLFIRI, mIFL
Description: as for outcome 1
Time Frame: every 6 weeks until disease progression
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + FOLFIRI: Bevacizumab + Irinotecan + infusional 5-FU/LV with (celecoxib or placebo)
- Bevacizumab + mIFL: Bevacizumab + Irinotecan + modified-bolus 5-FU/LV with (celecoxib or placebo)
Arm/Group | Bevacizumab + FOLFIRI | Bevacizumab + mIFL
Number analyzed (Participants) | 57 | 60
months | 11.17 [9.00 to 17.41] | 8.31 [6.31 to 11.63]
Statistical Analysis 1: Comparison: Bevacizumab + FOLFIRI vs Bevacizumab + mIFL; Test type: Superiority or Other; p = 0.2835, Log Rank; Hazard Ratio (HR) = 1.269, 95% CI [0.75 to 2.15]

10. Secondary Outcome: Overall Response: Bevacizumab With FOLFIRI, mIFL
Description: as for outcome 7
Time Frame: every 6 weeks during chemotherapy until disease progression
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + FOLFIRI | Bevacizumab + mIFL
Number analyzed (Participants) | 57 | 60
participants | 33 | 32
Statistical Analysis 1: Comparison: Bevacizumab + FOLFIRI; Test type: Superiority or Other; F-distribution method = 57.9, 95% CI [44.08 to 70.86] — Exact confidence interval for binomial proportion using the F-distribution method (unit: %)
Statistical Analysis 2: Comparison: Bevacizumab + mIFL; Test type: Superiority or Other; F-distribution method = 53.3, 95% CI [40.00 to 66.33] — Exact confidence interval for binomial proportion using the F-distribution method (unit: %)
Statistical Analysis 3: Comparison: Bevacizumab + FOLFIRI vs Bevacizumab + mIFL; Test type: Superiority or Other; p = 0.7388, Cochran-Mantel-Haenszel

11. Secondary Outcome: 1 Year Survival: Bevacizumab With FOLFIRI, mIFL
Description: as for outcome 5
Time Frame: 1 year from date of randomization
Population: ITT Population.
Measure: Number; unit: participants
Groups:
- Bevacizumab + mIRI: Bevacizumab + Irinotecan + modified-bolus 5-FU/LV with (celecoxib or placebo)
Arm/Group | Bevacizumab + FOLFIRI | Bevacizumab + mIRI
Number analyzed (Participants) | 57 | 60
participants
  Alive at 1 year | 45 | 33
  Dead at 1 year | 7 | 22
  Censored | 5 | 5

12. Secondary Outcome: Survival Time at Last Follow-Up Visit: Bevacizumab With FOLFIRI, mIFL
Description: Survival time defined as time from date of randomization to date of death. In the absence of confirmation of death, survival time was censored to last date the subject known to be alive. Zero subjects analyzed indicates median could not be analyzed based on number of subjects who died.
Time Frame: Last Follow-Up Visit
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + FOLFIRI | Bevacizumab + mIRI
Number analyzed (Participants) | 57 | 60
months | 27.99 [23.82 to 34.76] | 19.22 [11.60 to 22.28]
Statistical Analysis 1: Comparison: Bevacizumab + FOLFIRI vs Bevacizumab + mIRI; Test type: Superiority or Other; p = 0.0370, Log Rank; Hazard Ratio (HR) = 1.794, 95% CI [1.12 to 2.88]

13. Secondary Outcome: Dose Reduction Due to Treatment Emergent Adverse Events
Description: Number of subjects that had at least one Treatment-Emergent Adverse Event (TEAE) that led to a dose reduction. TEAE includes all reported Adverse Events that occurred within 30 days of last study medication.
Time Frame: Day 1; Day 8; and at end of every 3 treatment cycles for FOLFIRI; end of every 2 cycles for mIRI
Population: As-Treated population - all subjects who received any study medication, with treatment assignments designated according to actual study treatment received.
Measure: Number; unit: participants
Arm/Group | FOLFIRI | mIFL | CapeIRI | Bevacizumab + FOLFIRI | Bevacizumab + mIRI
Number analyzed (Participants) | 137 | 137 | 141 | 56 | 59
participants | 18 | 14 | 39 | 6 | 8

14. Secondary Outcome: Overall Relative Dose Intensity of Irinotecan
Description: Relative dose intensity for a cycle was calculated as the percentage of the actual dose intensity of the cycle divided by the planned dose intensity of the cycle. Overall relative dose intensity was calculated as the average relative dose intensities over all cycles. (Dose intensity for each cycle was calculated as the actual dose level of the study medication received in that cycle divided by the number of weeks in the cycle.)
Time Frame: End of treatment cycle
Population: As-Treated population
Measure: Mean (Standard Error); unit: percent dose intensity
Arm/Group | FOLFIRI | mIFL | CapeIRI | Bevacizumab + FOLFIRI | Bevacizumab + mIRI
Number analyzed (Participants) | 137 | 137 | 145 | 56 | 59
percent dose intensity | 93.9 (0.6) | 94.5 (0.6) | 93.8 (0.7) | 93.3 (0.8) | 95.5 (0.8)

ADVERSE EVENTS:
Arm/Group | FOLFIRI | mIFL | CapeIRI | Bevacizumab + FOLFIRI | Bevacizumab + mIRI
Serious Adverse Events (participants affected / at risk) | 50/137 | 52/137 | 78/141 | 19/56 | 21/59
Other Adverse Events (participants affected / at risk) | 135/137 | 137/137 | 140/141 | 56/56 | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI (N=137) | mIFL (N=137) | CapeIRI (N=141) | Bevacizumab + FOLFIRI (N=56) | Bevacizumab + mIRI (N=59)
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 12 | 8 | 3 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 4 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 6 | 5 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 8 | 42 | 2 | 4
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 5 | 2 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 20 | 5 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 3 | 7 | 2 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 6 | 24 | 5 | 2
Asthenia (General disorders) | 0 | 2 | 2 | 0 | 1
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 1 | 2 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 5 | 4 | 2 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Central line infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1 | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Polytraumatism (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Culture stool positive (Investigations) | 0 | 2 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 0 | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 7 | 24 | 4 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 3 | 0 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 8 | 2 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 5 | 4 | 2 | 1
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 2 | 0 | 0 | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Urinoma (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI (N=137) | mIFL (N=137) | CapeIRI (N=141) | Bevacizumab + FOLFIRI (N=56) | Bevacizumab + mIRI (N=59)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 17 | 10 | 3 | 1
Vertigo (Ear and labyrinth disorders) | 8 | 3 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 12 | 4 | 16 | 7 | 3
Vision blurred (Eye disorders) | 7 | 5 | 7 | 1 | 4
Abdominal discomfort (Gastrointestinal disorders) | 7 | 2 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 11 | 7 | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 65 | 50 | 61 | 20 | 18
Abdominal pain lower (Gastrointestinal disorders) | 0 | 7 | 5 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 15 | 12 | 14 | 9 | 7
Constipation (Gastrointestinal disorders) | 47 | 48 | 36 | 28 | 22
Diarrhoea (Gastrointestinal disorders) | 103 | 107 | 126 | 45 | 46
Dyspepsia (Gastrointestinal disorders) | 24 | 21 | 21 | 7 | 11
Flatulence (Gastrointestinal disorders) | 16 | 14 | 13 | 7 | 2
Haemorrhoids (Gastrointestinal disorders) | 9 | 4 | 5 | 6 | 7
Nausea (Gastrointestinal disorders) | 104 | 93 | 108 | 46 | 37
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 8 | 7 | 5 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 3 | 8 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 52 | 42 | 33 | 27 | 12
Vomiting (Gastrointestinal disorders) | 59 | 61 | 84 | 37 | 16
Asthenia (General disorders) | 18 | 17 | 23 | 6 | 7
Chest pain (General disorders) | 10 | 3 | 8 | 6 | 4
Chills (General disorders) | 12 | 14 | 12 | 8 | 3
Fatigue (General disorders) | 107 | 95 | 82 | 43 | 37
Mucosal inflammation (General disorders) | 19 | 13 | 14 | 12 | 6
Oedema (General disorders) | 8 | 6 | 6 | 0 | 0
Oedema peripheral (General disorders) | 23 | 18 | 24 | 5 | 2
Pyrexia (General disorders) | 30 | 28 | 28 | 12 | 6
Herpes simplex (Infections and infestations) | 8 | 6 | 5 | 0 | 0
Infection (Infections and infestations) | 3 | 8 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 8 | 4 | 2 | 3
Rhinitis (Infections and infestations) | 5 | 7 | 5 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 9 | 5 | 5 | 3
Urinary tract infection (Infections and infestations) | 4 | 9 | 6 | 6 | 3
Weight decreased (Investigations) | 10 | 12 | 15 | 5 | 4
Weight increased (Investigations) | 12 | 9 | 5 | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 41 | 42 | 48 | 22 | 17
Dehydration (Metabolism and nutrition disorders) | 24 | 18 | 42 | 9 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 19 | 10 | 12 | 10 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 8 | 19 | 11 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 8 | 6 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 16 | 13 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 13 | 11 | 13 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 3 | 4 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 8 | 4 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 3 | 7 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 7 | 6 | 3 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 12 | 13 | 7 | 3
Dizziness (Nervous system disorders) | 26 | 19 | 12 | 17 | 4
Dysgeusia (Nervous system disorders) | 22 | 20 | 20 | 10 | 3
Headache (Nervous system disorders) | 27 | 24 | 14 | 17 | 9
Hypoaesthesia (Nervous system disorders) | 7 | 3 | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 5 | 5 | 5 | 3
Syncope (Nervous system disorders) | 7 | 3 | 4 | 0 | 0
Anxiety (Psychiatric disorders) | 15 | 6 | 10 | 7 | 6
Confusional state (Psychiatric disorders) | 5 | 5 | 7 | 3 | 1
Depression (Psychiatric disorders) | 16 | 14 | 16 | 8 | 6
Insomnia (Psychiatric disorders) | 32 | 31 | 19 | 15 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 15 | 15 | 19 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 19 | 16 | 10 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 | 14 | 2 | 21 | 16
Hiccups (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 8 | 5 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 6 | 5 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 6 | 9 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 8 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 4 | 6 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 64 | 57 | 61 | 21 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 7 | 6 | 13 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 | 8 | 9 | 2 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 | 7 | 67 | 12 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 5 | 6 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 20 | 17 | 22 | 16 | 7
Deep vein thrombosis (Vascular disorders) | 17 | 11 | 11 | 5 | 2
Flushing (Vascular disorders) | 15 | 5 | 4 | 3 | 2
Hot flush (Vascular disorders) | 10 | 5 | 5 | 5 | 4
Hypertension (Vascular disorders) | 7 | 3 | 3 | 12 | 12
Hypotension (Vascular disorders) | 8 | 6 | 7 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 6 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 7 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 6
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 5
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3
Chest discomfort (General disorders) | 0 | 0 | 0 | 3 | 0
Malaise (General disorders) | 0 | 0 | 0 | 4 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 3 | 1
Pain (General disorders) | 0 | 0 | 0 | 3 | 2
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 4 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 6
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 3 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 6 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 3
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 7 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 3
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 3
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other